CLINICAL TRIAL: NCT07227727
Title: Endothelial Dysfunction After SCI: Mechanism and Therapeutic Target for SCI-related Cardiovascular Disease
Brief Title: Endothelial Dysfunction After SCI
Acronym: EDASCI
Status: Recruiting | Type: Observational
Sponsor: Craig Hospital (Other)
Collaborators: University of Colorado, Boulder (Other); Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Andrew Park, Physician Researcher at Craig Hospital, Craig Hospital
Other Study IDs: 1341523; 1341523 (Other Grant/Funding Number: Craig H Neilsen Foundation)
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Endothelial Dysfunction
Keywords: spinal cord injury; endothelium-dependent vasodilation; extracellular vesicles; microvesicles
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Cord Injury: Willing and eligible adults over the age of 18 years who sustained a motor complete (AIS A/B) paraplegia (neurological level of injury at T2 or below) spinal cord injury greater than 12 months ago. Participants of all races and ethnic backgrounds will be included in this study.
  Interventions: Procedure: Intra-arterial Infusion of Vasoactive Agents; Procedure: Intra-arterial Vitamin C Infusion; Procedure: Blood Sampling
- Control (Non-Spinal Cord Injury): Adults greater than 18 years of age who have never sustained a spinal cord injury. Participants of all races and ethnic backgrounds will be included in this study
  Interventions: Procedure: Intra-arterial Infusion of Vasoactive Agents; Procedure: Intra-arterial Vitamin C Infusion; Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Intra-arterial Infusion of Vasoactive Agents — A catheter is placed in the brachial artery of the non-dominant arm, and small doses of vasoactive drugs [acetylcholine (Ach), isoproterenol (ISO), sodium nitroprusside (SNP)] are infused. Forearm blood flow (FBF) is measured using venous occlusion plethysmography. The purpose of this procedure is to assess endothelium-dependent and independent vasodilation by stimulating different vascular pathways. The Ach infusion is to test muscarinic receptor, nitro oxide (NO) dependent, endothelium-dependent vasodilation. ISO infusion is to evaluate β-adrenergic, NO-dependent endothelium-dependent vasodilation. SNP infusion is to assess endothelium-independent vasodilation.
Procedure: Intra-arterial Vitamin C Infusion — Vitamin C, a potent antioxidant, will be infused into the arm and forearm blood flow (FBF) will be re-evaluated to determine whether oxidative stress contributes to endothelial dysfunction.
Procedure: Blood Sampling — Blood will be sampled from the antecubital vein (~50 mL) for biomarker analysis. This is to assess circulating biochemical and molecular indicators of vascular health and inflammation including levels of endothelial cell derived microvesicles (EMVs)

SUMMARY:
This study plans to learn how endothelial cells, single cell lining of blood vessels may be dysfunctional after a spinal cord injury. Endothelial dysfunction will be measured by the capacity of blood vessels to vasodilate (increase in size) and alter blood flow is lower in adults with a spinal cord injury in comparison to adults without a spinal cord injury. The mechanisms which may alter this function may be critical in reducing the risk of heart attacks and strokes in people with spinal cord injuries.

DETAILED DESCRIPTION:
Vascular endothelial dysfunction is prevalent after spinal cord injury (SCI) which predispose individuals with SCI to accelerated, atherosclerotic cardiovascular disease (ASCVD) and future myocardial infarctions and ischemic strokes. The central objective of this study is to determine whether adults with SCI exhibit impaired endothelial function. Specifically, if endothelium-dependent vasodilation is impaired and if endothelial cell derived microvesicles (EMVs) are elevated and dysfunctional in adults with paraplegia. Endothelium-dependent vasodilation will be assessed by pharmacologically manipulating endothelial vasodilator function in live conscious humans with SCI and determining the role of circulating EMVs as both a systemic biomarker and mediator of endothelial dysfunction.

ELIGIBILITY:
SCI Inclusion Criteria

* Over age 18 years
* Chronic (>12 months) SCI
* Motor complete (AIS A/B) SCI
* Paraplegia (neurological level of injury [NLI] at T2 or below)

Non-injured Inclusion Criteria

• Over age 18 years

Exclusion Criteria (Both SCI and Non-injured)

* Overt chronic diseases as assessed by: a) clinically documented medical history; b) physical examination; c) blood pressure and ECG at rest; and d) complete blood chemistries and hematological evaluation.
* Active infection
* Recent (< 3 months) surgery
* Current smoking history (within past 12 months)
* Report more than low-risk alcohol consumption
* History of drug abuse
* Currently taking cardiovascular (statins, beta-blockers) therapeutics and/or other medications that could influence the outcome measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants of this study will all be willing and eligible adults who sustained a spinal cord injury, and adults who have never sustained a spinal cord injury. Participants of all races and ethnic backgrounds will be included in this study. A total up to 40 participants will be enrolled with the goal of 20 in each group to complete the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Endothelium-dependent vasodilation | Measured at baseline and immediately after each vasoactive dose for 3-5 minutes.
  Total forearm blood flow with be measured by strain gauge venous plethysmography under baseline conditions and under pharmacological manipulation with acetylcholine and isoproterenol at increasing concentrations.
Endothelium-independent vasodilation | Measured at baseline (without sodium nitroprusside) and immediately after each sodium nitroprusside dose for 3-5 minutes.
  Total forearm blood flow with be measured by strain gauge venous plethysmography under baseline conditions and under pharmacological manipulation with sodium nitroprusside at increasing concentrations (1, 2, 4ug/ml).
Endothelial cell-derived microvesicles concentration | Baseline
  Endothelial cell-derived microvesicles will be collected from venous blood samples and counted used flow cytometry to determine a circulating concentration.
Endothelial cell-derived microvesicles effects of human coronary artery endothelial cells nitric oxide bioavailability | Baseline
  Endothelial cell-derived microvesicles will be sorted and collected by fluorescence-activated cell sorting (FACS) flow cytometry. The endothelial cell-derived microvesicles will be co-cultured with human coronary artery endothelial cells. Endothelial Nitric Oxide Synthase and phosphorylation sites of interest will be measured by intracellular protein expression quantification of whole cell lysates by capillary electrophoresis immunoassays. Nitric oxide production will be assessed by total nitric oxide and nitrate/nitrite parameter assays.
Endothelial cell-derived microvesicles effects of human coronary artery endothelial cells reactive oxygen species and antioxidant capacity | Baseline
  Endothelial cell-derived microvesicles will be sorted and collected by fluorescence-activated cell sorting (FACS) flow cytometry. The endothelial cell-derived microvesicles will be co-cultured with human coronary artery endothelial cells. Super oxide dismutase and catalase expression will be measured by intracellular protein expression quantification of whole cell lysates by capillary electrophoresis immunoassays. Intracellular oxidative stress will be assessed by ROS-Glo H2O2 assay.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Park, MD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be facilitated through active participation in Open Data Commons for SCI (ODC-SCI). ODC-SCI is a cloud-based community-governed repository to store, share, and publish research data on Spinal Cord Injury and is compliant with requirements for FAIR and trustworthy repositories established by NIH.